CLINICAL TRIAL: NCT04265742
Title: Microbiota and Bone Fragility: Study of the Relation Between Gut Microbiota and Bone Microarchitecture (Microbone)
Brief Title: Microbiota and Bone Fragility:Study of the Relation Between Gut Microbiota and Bone Microarchitecture
Acronym: MICROBONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: C18-04; 2018-A01806-49 (Registry Identifier: MICROBONE)
Record Dates: First submitted 2018-09-24; First posted 2020-02-12 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2021-08

CONDITIONS: Bone Loss, Age-related
Keywords: Bone microarchitecture; intestinal microbiote; post-menopausal women; bone remodeling
MeSH Terms: conditions — Osteoporosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: The composition of the intestinal microbiota will be evaluated by the ratio between the amount of pro-inflammatory bacteria (Prevotellaceae, E. coli, Bacteroides vulgatus, Proteus mirabili) and the amount of anti-inflammatory bacteria (Faecalibacterium, Roseburia) in postmenopausal women with comparable bone mineral density, according to their fracture status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A. Normal BMD, no fracture (Experimental): Post-menopausal women with normal bone density (BMD t-score >-1.5) and no history of fractures. Intervention: bone densitometry, high resolution peripheral QCT(HR-pQCT), collection of biological samples, questionnaires, clinical tests.
  Interventions: Radiation: bone densitometry; Radiation: High resolution peripheral QCT; Diagnostic Test: Collection of biological samples; Other: questionnaires; Other: clinical tests
- Group B. Normal BMD, with fracture (Experimental): Post-menopausal women with normal bone density (BMD T-score >-1.5) with history of fractures. Intervention: bone densitometry, high resolution peripheral QCT(HR-pQCT), collection of biological samples, questionnaires, clinical tests.
  Interventions: Radiation: bone densitometry; Radiation: High resolution peripheral QCT; Diagnostic Test: Collection of biological samples; Other: questionnaires; Other: clinical tests
- Group C. osteoporotic, no fracture (Experimental): Post-menopausal women with low bone density (BMD T-score <-2.5) and no history of fractures. Intervention: bone densitometry, high resolution peripheral QCT(HR-pQCT), collection of biological samples, questionnaires, clinical tests.
  Interventions: Radiation: bone densitometry; Radiation: High resolution peripheral QCT; Diagnostic Test: Collection of biological samples; Other: questionnaires; Other: clinical tests
- Group D. osteoporotic, with fracture (Experimental): Post-menopausal women with low bone density (BMD T-score <-2.5) with history of fractures. Intervention: bone densitometry, high resolution peripheral QCT(HR-pQCT), collection of biological samples, questionnaires, clinical tests.
  Interventions: Radiation: bone densitometry; Radiation: High resolution peripheral QCT; Diagnostic Test: Collection of biological samples; Other: questionnaires; Other: clinical tests

INTERVENTIONS:
Radiation: bone densitometry — Bone Mineral Density (BMD), body composition, vertebral fractures
Radiation: High resolution peripheral QCT — High resolution peripheral QCT (HR-pQCT): bone microarchitecture and bone strength
Diagnostic Test: Collection of biological samples — Peripheral blood and urine samples to assess bone turnover markers and cytokines; and faeces to assess gut microbiota composition
Other: questionnaires — Epidemiologic and nutritional questionnaire and physical activity scale
Other: clinical tests — physical performance tests and grip strenght measurement

SUMMARY:
Gut microbiota regulate metabolism of their human host. Some diseases are associated with variations in gut microbiota diversity and higher fracture risk. Intestinal bacteria synthesize or influence synthesis of factors modulating bone metabolism. The link between gut microbiota and bone was assessed mainly in experimental animal studies. Clinical data, e.g. on the role of gut microbiota in postmenopausal osteoporosis are scarce. The investigators will compare gut microbiota composition in four groups of women aged ≥60 recruited on the basis of bone mineral density (BMD) and personal history of fracture. the participants will have diagnostic exams: clinical tests, bone densitometry (body composition, vertebral fractures), high resolution peripheral QCT (bone strength estimated by microfinite element analysis, micro-FEA), biological sample collection. Gut microbiome profiling will be performed at the INRA MetaGenoPolis laboratory. The investigators will compare gut microbiota diversity according to BMD level and to the fracture status. The investigators will analyze interactions of the gut microbiota diversity with bone status (bone turnover rate, BMD, bone microarchitecture, bone strength estimated by micro-FEA), muscle mass and strength, inflammatory cytokines and micro-RNAs modulating their expression. This study will provide new data concerning the importance of gut microbiota for the fracture risk in older women. It will help to identify the main metabolic pathways underlying the observed associations.

DETAILED DESCRIPTION:
Postmenopausal osteoporosis is a major public health problem in developed countries. Despite the progress, knowledge of its pathophysiological mechanisms and identification of women at high risk of fracture in the clinical practice are not satisfactory. Gut microbiota consist of trillions of commensal bacteria playing a major role in the regulation of metabolism of their human host. Some conditions (diabetes mellitus, obesity, liver cirrhosis, inflammatory bowel disease, end stage renal disease, depression, heavy drinking, heavy smoking) are associated with variations in gut microbiota diversity and higher risk of fracture. Intestinal bacteria synthesize or influence the synthesis of factors which modulate bone metabolism, e.g. lipopolysaccharide (present in the wall of Gram-negative bacteria), inflammatory cytokines (synthesized in the gut associated lymphoid tissue), serotonin (synthesized in the colon epithelium), short-chain fatty acids, estrogens (deconjugation of sulphates and glucuronides). Data on the association between gut microbiota and bone metabolism were obtained mainly in experimental animal studies. Clinical data are limited. Data on the possible role of gut microbiota in the pathophysiology of the postmenopausal osteoporosis are scarce.

The investigators will carry out a cross-sectional comparison of gut microbiota composition in four groups of women aged 60 and over recruited on the basis of their bone mineral density (BMD) and personal history of fragility fracture. The primary statistical analyses will be focused on the comparison of gut microbiota diversity according to BMD (in women with the same fracture status) and according to the fracture status (in women with similar BMD). The investigators will analyze interactions of the gut microbiota diversity, its metabolic activity and other metabolic factors on the one hand, with bone status on the other hand. The investigators will study the association of gut microbiota composition with bone turnover rate, BMD, bone microarchitecture, bone strength estimated by microfinite element analysis (micro-FEA) and with physical performance, muscle mass and strength. The investigators will assess the impact of microRNAs modulating the expression of inflammatory cytokines on the serum levels of these cytokines according to the pattern of gut microbiota diversity and their associations with the characteristics of bone status (e.g. bone microarchitecture). The investigators will analyze the association between serum serotonin, abundance of intestinal bacteria stimulating serotonin synthesis (some Clostridia species) in the colon and the characteristics of bone status.

This study will provide new data concerning the importance of gut microbiota for the fracture risk in older women. The main limitation of this study is its cross-sectional design but this is the first clinical study exploring this subject. It will help to identify the main metabolic pathways underlying the observed associations. These data will stimulate experimental studies to elucidate biological mechanisms underlying these associations. the results will provide indications for future clinical and experimental studies. In the long run, the results will lead up to future studies permitting to develop new biological markers of fracture risk in older women and new anti-osteoporotic medications.

ELIGIBILITY:
Inclusion Criteria:

* post-menopausal women
* with a normal Bone Mineral Density (T-score >-1.5) at the 3 sites (lumbar spine, total hip and femoral neck) or with osteoporosis (T-score ≤ -2.5) at least at one of the 3 sites.

Exclusion Criteria:

* Current antibiotherapy or in the last 6 months or repeated antibiotherapy
* Current corticotherapy or stopped for less than 6 months
* Current treatment of osteoporosis or having lasted more than 3 months in the last 5 years
* Current hormonal treatment for menopause
* Current or discontinued drugs that may affect bone metabolism (eg anti-aromatase)
* Known hepatic, cardiac or respiratory insufficiency
* Pathologies that may affect bone metabolism, particularly severe renal insufficiency
* Serious illnesses, particularly disabling and chronic diseases of the gastrointestinal tract
* Diseases characterized by substantial disorders of the gut microbiota (eg severe obesity, BMI> 40 kg / m2, depression, poorly controlled diabetes)
* Psychiatric pathology hindering understanding
* Difficulty understanding oral French
* Person protected by law, unable to express her consent, subject to a protective measure or deprived of liberty.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
Comparison of the composition of the gut microbiota according to fracture status in postmenopausal women with comparable bone mineral density. | through study completion, an average of 3 years
  The composition of the intestinal microbiota will be evaluated by the ratio between the amount of proinflammatory bacteria (Prevotellaceae, E. coli, Bacteroides vulgatus, Proteus mirabili) and the amount of anti-inflammatory bacteria (Faecalibacterium, Roseburia) in postmenopausal women with mineral density comparable bone according to their fracture status.

SECONDARY OUTCOMES:
Determine the relationship between the composition of the gut microbiota and bone microarchitecture according to fracture status in postmenopausal women with comparable bone mineral density. | through study completion, an average of 3 years
  Relationship between gut microbiota composition (evaluated by the ratio between the amount of proinflammatory bacteria (Prevotellaceae, E. coli, Bacteroides vulgatus, Proteus mirabili) and the amount of anti-inflammatory bacteria (Faecalibacterium, Roseburia)) and bone microarchitecture of the distal radius and tibia measured by High resolution peripheral QCT in each of the 4 groups of women (Normal BMD with or without fracture, osteoporosis with or without fracture).
Determine the relationship between the composition of the gut microbiota and bone mineral density according to fracture status in postmenopausal women with comparable bone mineral density. | through study completion, an average of 3 years
  Relationship between gut microbiota composition (evaluated by the ratio between the amount of proinflammatory bacteria (Prevotellaceae, E. coli, Bacteroides vulgatus, Proteus mirabili) and the amount of anti-inflammatory bacteria (Faecalibacterium, Roseburia)) and bone mineral density measured by DXA in each of the 4 groups of women (Normal BMD with or without fracture, osteoporosis with or without fracture).
Determine the relationship between the composition of the gut microbiota and muscle mass and strength according to fracture status in postmenopausal women with comparable bone mineral density. | through study completion, an average of 3 years
  Relationship between gut microbiota composition (evaluated by the ratio between the amount of proinflammatory bacteria (Prevotellaceae, E. coli, Bacteroides vulgatus, Proteus mirabili) and the amount of anti-inflammatory bacteria (Faecalibacterium, Roseburia)) and muscle mass (assessed by whole body composition measured by DXA) and strength (assessed by dynamometry) in each of the 4 groups of women (Normal BMD with or without fracture, osteoporosis with or without fracture).
Determine the relationship between the composition of the gut microbiota and physical performance according to fracture status in postmenopausal women with comparable bone mineral density. | through study completion, an average of 3 years
  Relationship between gut microbiota composition (evaluated by the ratio between the amount of proinflammatory bacteria (Prevotellaceae, E. coli, Bacteroides vulgatus, Proteus mirabili) and the amount of anti-inflammatory bacteria (Faecalibacterium, Roseburia)) and physical performance (assessed by gait speed and clinical tests) in each of the 4 groups of women (Normal BMD with or without fracture, osteoporosis with or without fracture).
Determine the relationship between the composition of the gut microbiota and bone remodeling according to fracture status in postmenopausal women with comparable bone mineral density. | through study completion, an average of 3 years
  Relationship between gut microbiota composition( evaluated by the ratio between the amount of proinflammatory bacteria (Prevotellaceae, E. coli, Bacteroides vulgatus, Proteus mirabili) and the amount of anti-inflammatory bacteria (Faecalibacterium, Roseburia)) and bone remodeling (evaluated by biochemical bone remodeling markers) in each of the 4 groups of women (Normal BMD with or without fracture, osteoporosis with or without fracture).
Determine the relationship between the composition of the gut microbiota and regulatory hormones of bone metabolism according to fracture status in postmenopausal women with comparable bone mineral density. | through study completion, an average of 3 years
  Relationship between gut microbiota composition (evaluated by the ratio between the amount of proinflammatory bacteria (Prevotellaceae, E. coli, Bacteroides vulgatus, Proteus mirabili)) and the amount of anti-inflammatory bacteria (Faecalibacterium, Roseburia) and regulatory hormones of bone metabolism (measured by dosages) in each of the 4 groups of women (Normal BMD with or without fracture, osteoporosis with or without fracture).
Determine the relationship between the composition of the gut microbiota and genetic factors according to fracture status in postmenopausal women with comparable bone mineral density. | through study completion, an average of 3 years
  Relationship between gut microbiota composition (evaluated by the ratio between the amount of proinflammatory bacteria (Prevotellaceae, E. coli, Bacteroides vulgatus, Proteus mirabili) and the amount of anti-inflammatory bacteria (Faecalibacterium, Roseburia)) and genetic regulation assessed by GWAS (genome-wide association study) and miRNA study in each of the 4 groups of women (Normal BMD with or without fracture, osteoporosis with or without fracture).

CONTACTS AND LOCATIONS:
Overall Officials: Pawel SZULC, MD, Ph.D, Principal Investigator — Hospital Edouard Herriot, , 69437 Lyon
Locations (1):
- Hopital E. Herriot, Lyon, France